CLINICAL TRIAL: NCT03749850
Title: Image-guided Targeted Doxorubicin Delivery With Hyperthermia to Optimize Loco-regional Control in Breast Cancer. Phase I Feasibility Study of Hifu-Induced Hyperthermia, LTLD and Cyclophosphamide for Metastatic Breast Cancer
Brief Title: Image-guided Targeted Doxorubicin Delivery With Hyperthermia to Optimize Loco-regional Control in Breast Cancer
Acronym: i-GO
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Dutch Cancer Society (Other); Center for Translational Molecular Medicine (Other); Vrienden UMC Utrecht (Unknown)
Responsible Party: Principal Investigator, BBM Suelmann, Principal Investigator, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL67422.041.18; 2015-005582-23 (EudraCT Number)
Record Dates: First submitted 2018-11-09; First posted 2018-11-21 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Metastatic Breast Cancer; Breast Cancer; Breast Neoplasms; Stage IV Breast Cancer; Metastatic Cancer; Invasive Ductal Carcinoma of Female Breast; Invasive Ductal Breast Cancer; Adenocarcinoma Breast
Keywords: High Intensity Focused Ultrasound; lyso-thermosensitive liposomal doxorubicin; ThermoDox; MR-HIFU; mild local hyperthermia; local drug delivery; image-guided therapy; nanomedicine; liposome; doxorubicin; adriamycin; cyclophosphamide; HIFU; LTLD; hyperthermia; de novo stage IV; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Carcinoma, Ductal, Breast; Hyperthermia | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study treatment (Experimental): LTLD in combination with MR-HIFU induced hyperthermia and cyclophosphamide
  Single arm study
  Interventions: Drug: LTLD; Procedure: MR-HIFU induced hyperthermia; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: LTLD — Patients will receive up to six cycles at three-weeks intervals of:
  * Intravenous LTLD dosed at 50mg/m2 administered during the MR-HIFU treatment
  * 60 minutes of MR-HIFU mild local hyperthermia at 40 °C - 42 °C to the primary breast tumour
  * Intravenous Cyclophosphamide 600 mg/m2 after MR-HIFU treatment
  In case of toxicity, LTLD, cyclophosphamide and/or hyperthermia dosages will be adjusted as specified in the study protocol.
  Other Names: ThermoDox; Lyso-Thermosensitive Liposomal Doxorubicin
Procedure: MR-HIFU induced hyperthermia — Patients will receive up to six cycles at three-weeks intervals of:
  - 60 minutes of MR-HIFU mild local hyperthermia at 40 °C - 42 °C to the primary breast tumour.
  In case of toxicity, hyperthermia dosages will be adjusted as specified in the study protocol.
  Other Names: MR-HIFU; Magnetic Resonance guided High Intensity Focused Ultrasound; MLHT; Mild local hyperthermia
Drug: Cyclophosphamide — Patients will receive up to six cycles at three-weeks intervals of:
  - Intravenous Cyclophosphamide 600 mg/m2 after MR-HIFU treatment
  In case of toxicity, cyclophosphamide dosages will be adjusted as specified in the study protocol.
  Other Names: Endoxan

SUMMARY:
In this phase I feasibility study, the investigators evaluate the combination of lyso-thermosensitive liposomal doxorubicin (LTLD, ThermoDox) with local hyperthermia and cyclophosphamide (C), for the local treatment of the primary breast tumour in patients with metastatic breast cancer.

When heated to 40-43 degrees Celsius (ºC), LTLD releases a very high concentration of doxorubicin locally within seconds. Hyperthermia of the primary tumour will be induced by Magnetic Resonance guided High Intensity Focused Ultrasound (MR-HIFU) on a dedicated Sonalleve MR-HIFU breast system.

The investigators hypothesize that by substituting doxorubicin (A) in the AC-chemotherapy regimen for the combination of LTLD and MR-HIFU induced hyperthermia, optimal local tumour control can be achieved without compromising systemic toxicity or efficacy.

This will be the first study to evaluate LTLD with MR-HIFU hyperthermia in breast cancer patients.

DETAILED DESCRIPTION:
Advances in systemic treatment led to improved overall survival in patients with metastatic breast cancer. Various studies suggest that by obtaining loco-regional control, overall survival in advanced disease can further be improved.

Pre-operative chemotherapy can be used in metastatic breast cancer to make radical removal of the primary tumor feasible, while simultaneously maintaining control of already present metastatic sites. The doxorubicin and cyclophosphamide regimen (AC) is well-known both in (neo-)adjuvant setting as in treatment of metastatic breast cancer. At present, optimal local control in advanced breast cancer using adequate dosing of doxorubicin is hampered by its toxic systemic effects. Therefore the investigators aim to increase doxorubicin deposition in the primary tumor without interfering with systemic efficacy and toxicity, by combining lyso-thermosensitive liposomal doxorubicin (LTLD, ThermoDox) with local mild hyperthermia, induced by Magnetic Resonance guided High Intensity Focused Ultrasound (MR-HIFU). When heated to 40-43 ºC, ThermoDox releases a very high concentration of doxorubicin locally within seconds. In the absence of hyperthermia, ThermoDox leads to a similar biodistribution and antitumor efficacy to free doxorubicin. MR-HIFU allows for controlled heating of deep-seated tumors.

This is a single-arm phase I feasibility study in 12 patients with de novo stage IV (distant metastasis at the time of diagnosis) her2-negative breast cancer, who have not received previous chemotherapy. The study treatment consists of up to 6 cycles at 21-day intervals of ThermoDox (50mg/m2) administered during MR-HIFU induced hyperthermia (60 minutes at 40-42 ᵒC) and cyclophosphamide (600 mg/m2) administered afterwards. A dedicated MR-HIFU breast system integrated with a clinical 1.5 Tesla Magnetic Resonance Imaging (MRI) scanner will be used for safe and controlled heating of the tumour. Primary endpoints are safety, tolerability and feasibility. Secondary endpoint is efficacy, assessed by radiological response of the local tumor and the distant metastases.

In the Biobank side study, extra blood samples will be collected. These samples will be used for further research on not yet determined topics related to breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria:

1. Histologically confirmed adenocarcinoma of the breast and planned for palliative chemotherapy with doxorubicine en cyclophosphamide
2. Biopsy-proven stage tumor 1-2, any nodes, metastasis 1 (T1-2AnyNM1) at diagnosis of breast cancer.
3. Non-pregnant, non-lactating female at least 18 years of age. If patient is of child-bearing age, she must have a negative serum pregnancy test prior to enrollment and must agree to practice an acceptable form of birth control while on study.
4. The tumor is located within the reach of the HIFU beam (based on pre-treatment Dynamic Contrast Enhanced (DCE-) MRI findings).
5. The distance of the tumor from the skin, nipple, and pectoral wall is at least 1.0 cm (based on pre-treatment DCE-MRI findings).
6. The target breast is expected to fit in the cup of the dedicated MR-HIFU breast system (based on pre-treatment MRI findings).
7. The patient weighs less than 90 kg (restrictment of the HIFU table top).
8. Provide written informed consent and willing to comply with protocol requirements.

Exclusion Criteria:

Patients will be excluded if any of the following conditions are observed:

1. Her2-positive disease or classic invasive lobular carcinoma (ILC).
2. A treatment plan with curative intent is available.
3. Any prior chemotherapy treatment for invasive breast cancer (previous anti-hormonal therapy is allowed)
4. Any prior therapy with anthracyclines
5. No measurable disease at baseline (according to RECIST 1.1 or PERCIST 1.0)
6. Any concomitant malignancy or previous malignancy in the last 5 years, except basal cell or squamous cell cancer of the skin or in situ carcinoma of the cervix.

   Subjects with a prior contralateral breast malignancy more than 5 years ago can be included if they did not receive any chemotherapy.
7. Any previous malignancy in the unilateral breast (even if more than 5 years ago)
8. Prior sensitivity (including rash, dyspnea, wheezing, urticarial, or other symptoms) attributed to any liposomal-encapsulated drug.
9. Baseline laboratory values:

   Absolute Neutrophil Count (ANC) < 1.5 x 10^9/L, Platelets < 75 x 10^9/L, Hemoglobin < 5.6 mmol/L (9 g/dl), Total Bilirubin > 1.5 x upper limit of normal, Alanine Transaminase (ALAT) and Aspartate Transaminase (ASAT) > 2.5 x upper limit of normal >5 x upper limit of normal in case of liver metastases, Estimated Glomerular Filtration Rate (eGFR) < 30 ml/min/1.73m2.
10. World Health Organization Performance Status (WHO-PS) >2.
11. Left Ventricular Ejection Fraction <50% (validated by baseline scan).
12. History of:

    1. Acute coronary syndrome in the last year
    2. Cerebral vascular accident in the last year
    3. Abnormal cardiac stress testing within last 6 months
    4. Symptomatic coronary artery disease
    5. Uncontrolled hypertension or cardiomyopathy
    6. Cardiac valvular surgery or open heart surgery in the last year
    7. Known structural heart disease
13. Any condition which may interfere with the hyperthermia portion of the trial such as: functioning cardiac pacemaker; metal plates, rods or prosthesis of the chest wall, breast prosthesis in the treated breast, severe numbness and/or tingling of the chest wall or breast, skin grafts and/or flaps on the breast or chest wall, scar tissue or surgical clips in the HIFU beam path.
14. Active infection
15. Body temperature > 38.0 degrees Celsius on the day of a MR-HIFU treatment.
16. Concurrent use of any of the following prohibited medications within a reasonable wash-out time: protease inhibitors, cyclosporine, carbamazepine, phenytoin, valproic acid, paclitaxel, trastuzumab and other liposomal drugs (Abelect, Ambisome, Nyotran, etc.) or lipid-complexed drugs.
17. Caution will be exercised with all the medications mentioned in appendix C, for interactions are theoretically possible.
18. Contraindications to MR imaging (e.g., pacemaker in situ, severe claustrophobia, metal implants incompatible with the MRI-scan, body size incompatible with MR bore).
19. Contraindications to gadolinium-based contrast agent, including prior allergic reaction to gadolinium-based contrast agent, and/or renal failure.
20. Contraindications to sedation and analgesia with propofol and Remifentanil, including history of Chronic Obstructive Pulmonary Disease (COPD) that results in the inability to perform a physical activity corresponding with a Metabolic Equivalent (MET(57)) of 4; dependence on artificial ventilation at home; sleep apnea or an American Society of Anesthesiologists (ASA) classification ≥4.
21. Inability to lie in prone position.
22. A medical or psychiatric condition or other circumstances which would significantly decrease the chances of understanding the informed consent process, obtaining reliable data, achieving study objectives, or completing the study treatment and/or examinations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events assessed by CTCAE v 5.0 | From first study treatment (day 1) until the end of study visit between day 161 and 175
  Safety and tolerability of the study treatment
Incidence of dose limiting toxicities | From first study treatment (day 1) until the end of study visit between day 161 and 175
  Safety and tolerability of the study treatment
Incidence of necessity for dose adjustments, delay or early cessation | From first study treatment (day 1) until the end of study visit between day 161 and 175
  Safety and tolerability of the study treatment
Incidence and severity of post-procedural pain | From first study treatment (day 1) until the end of study visit between day 161 and 175
  Safety and tolerability of the study treatment
Patient reported tolerability via an adapted version of the Cancer Therapy Satisfaction Questionnaire (CTSQ) | Baseline, day 49 and day 112
  Tolerability of the study treatment. Scores will be described.
Patient reported tolerability via the Functional Assessment of Cancer Therapy - Breast (FACT-B) questionnaire | Baseline, and on day 14 of each cycle (with a maximum of six 21-day cycles in 18 weeks)
  Tolerability of the study treatment. Scores will be described.
Incidence of cardiotoxity | From first study treatment (day 1) until the end of study visit between day 161 and 175
  Safety and tolerability of the study treatment
Description of MR thermometry data (describing the temperatures achieved) | On day 1 (study treatment day) of each cycle (with a maximum of six 21-day cycles in 18 weeks)
  Feasibility of the study treatment
Duration of procedures on a treatment day | On day 1 (study treatment day) of each cycle (with a maximum of six 21-day cycles in 18 weeks)
  Feasibility of the study treatment
Number of completed cycles with MR-HIFU induced hyperthermia, ThermoDox and cyclophosphamide | From first study treatment (day 1) until the end of study visit between day 161 and 175
  Feasibility of the study treatment
The number of cycles in which hyperthermia was sufficient: at least 30 minutes at the target temperature of 40-42°C | From first study treatment (day 1) until the end of study visit between day 161 and 175
  Feasibility of the study treatment

SECONDARY OUTCOMES:
Radiological objective response locally on breast Magnetic Resonance Imaging, assessed by RECIST 1.1. | Assessed after 2 cycles and after 6 cycles of the study treatment. Each cycle is 21 days.
  Efficacy of the study treatment
Radiological objective response systemically on Computed Tomography, assessed by RECIST 1.1 or (for patients without RECIST-measurable disease) Positron Emission Tomography Computed Tomography, assessed by PERCIST 1.0 | Assessed after 2 cycles and after 6 cycles of the study treatment. Each cycle is 21 days.
  Efficacy of the study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Britt BM Suelmann, MD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Maar JS, Suelmann BBM, Braat MNGJA, van Diest PJ, Vaessen HHB, Witkamp AJ, Linn SC, Moonen CTW, van der Wall E, Deckers R. Phase I feasibility study of Magnetic Resonance guided High Intensity Focused Ultrasound-induced hyperthermia, Lyso-Thermosensitive Liposomal Doxorubicin and cyclophosphamide in de novo stage IV breast cancer patients: study protocol of the i-GO study. BMJ Open. 2020 Nov 26;10(11):e040162. doi: 10.1136/bmjopen-2020-040162. PMID 33243800